CLINICAL TRIAL: NCT06594614
Title: Observational Retrospective Study Describing Demographic, Clinical and Laboratory Characteristics and Survival Correlates of Progressive Multifocal Leukoencephalopathy (PML) in Italy, 1987-2024
Brief Title: Observational Study on Characteristics and Survival Correlates of Progressive Multifocal Leukoencephalopathy (PML) in Italy
Acronym: MI_PML
Status: Completed | Type: Observational
Sponsor: Scientific Institute San Raffaele (Other)
Responsible Party: Principal Investigator, Paola Cinque, Head of Clinical Research Unit, Scientific Institute San Raffaele
Other Study IDs: Milano PML cohort
Record Dates: First submitted 2024-09-10; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Progressive Multifocal Leukoencephalopathy; PML
Keywords: Progressive Multifocal Leukoencephalopathy; PML; epidemiology; survival; JCV-DNA; cerebrospinal fluid; JCV; JC virus; JC human polyomavirus; Human polyomavirus 2
MeSH Terms: conditions — Leukoencephalopathy, Progressive Multifocal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Cerebrospinal fluid, plasma, PBMCs
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with Progressive Multifocal Leukoencephalopathy

SUMMARY:
The goal of this observational study is to learn about the features of Progressive Multifocal Leukoencephalopathy (PML) at the time of its diagnosis and the factors that may influence the outcome of persons with this disease.

PML is a rare and rapidly progressive disease of the brain, caused by a virus named JC polyomavirus (JCV). This disease almost always occurs in persons with an immune dysfunction. In some people, the underlying immune dysfunction may be the consequence of other conditions, such as certain hematological tumors (for instance, some lymphomas) or the infection with the Human Immune Deficiency Virus (HIV). In other cases it may be associated with other forms of immune deficiency, either present at birth or acquired later in life, or with immunosuppressive or immunomodulant treatments, such as Natalizumab in persons with Multiple Sclerosis.

Unfortunately, there is no cure for PML, and the only possibility to stop the progression of the disease is to eliminate the cause of the underlying immune dysfunction. This is not always possible, or it may take time, and, therefore, more than half of the persons who developed PML will not survive to the disease.

This study takes advantage of the systematic collection, over a time frame of 37 years, of the characteristics of 456 cases of PML. The main question of this study aims to answer whether and how PML characteristics and outcome have evolved over time and also according to the disease or condition that caused the immune dysfunction leading to PML.

This is important because PML is a rare disease, and, therefore, knowing the context in which it develops can be useful for healthcare providers and families to consider PML as a possible cause of unexpected neurological problems. In fact, an early recognition of PML is associated with a better outcome. On the other hand, there are clinical and laboratory features of PML that can also be associated with different disease outcome. Therefore, it is important that these features are identified, to provide important information for disease management and also for the design of experimental therapeutic interventions.

Participants of this study are persons with a diagnosis of PML who were followed at the Infectious Diseases Unit of San Raffaele Hospital in Milan or referred to the Unit from other Italian clinical centers, between January 1st 1987 and April 30th 2024. We have retrospectively reviewed their clinical charts and collected demographic characteristics, together with the clinical, radiological and laboratory features of PML at the time of its diagnosis. In addition we have also reviewed the evolution of the disease one-year after the date of diagnosis.

The data from the participants have been collected in a custom-made database, which is kept updated with follow-up data and inclusion of new participants. As by April 30th 2024, 456 participants have been included in the database. This is one of the largest existing cohorts and the one with the longest observational window. In addition, and differently from previous cohort studies, it analyzes in detail clinical, radiological, and virological characteristics of PML, providing additional information on their changes over time and possible predictors of disease outcome.

DETAILED DESCRIPTION:
This is a retrospective observational study that investigates the features and the correlates of survival of patients with Progressive Multifocal Leukoencephalopathy (PML). The study is based on demographic, clinical and laboratory data stored in an Institutional database

PML is a rare and rapidly progressive demyelinating disease of the central nervous system (CNS), caused by the JC polyomavirus (JCV) that occurs in persons with a primary or acquired immune dysfunction. Common diseases or conditions associated with PML include certain hematological tumors (e.g., some lymphomas), Human Immune Deficiency Virus (HIV) infection, other congenital or acquired forms of immune deficiency, or in people receiving immunosuppressive or immunomodulant treatments, such as Natalizumab in persons with Multiple Sclerosis.

There is no specific effective treatment for PML, and reversion of the underlying immune dysfunction is the only feasible approach to halt disease progression. The overall reported mortality is higher than 50% and most of the persons who survive PML are left with severe neurological sequelae

Being PML a rare disease, knowing the context and the risk factors in which it develops, e.g., specific underlying diseases or treatments and their role in the different time periods, will be key for an early diagnosis of PML, which is usually associated with better outcome. In addition, the identification of variables associated with different disease outcomes will be important in terms of disease management and for the design of experimental therapeutic interventions.

The retrospective assessment of the PML cohort describes and analyzes clinical and laboratory data from 456 PML patients observed in the period 1987-2024. This is one of the largest cohorts and the with the longest observational window ever reported, reflecting an evolving epidemiological context. In addition, differently from previous cohort studies, it analyzes in detail clinical, radiological, and virological variables, providing additional information on the epidemiological changes and determinants of survival.

The cohort includes Italian PML patients who were followed at or referred to the Infectious Diseases Unit of San Raffaele Hospital in Milano, Italy from other Italian clinical centers, between January 1st 1987 and April 30th 2024. Data have been collected in a custom-made database, which is kept updated with follow-up data of cases already included and with inclusion of new cases. We have collected the demographic characteristics and the clinical, radiological and laboratory variables at first observation and at the time of diagnosis and at all the subsequent evaluations until death or up to three years in patients who survive.

More in detail, the following variables have been evaluated for the purpose of this study at the time of PML diagnosis: age, birth sex, year of diagnosis of PML, underlying PML disease, neurological deficits (classified as by presence of motor, cognitive, cerebellar, visual, verbal or cranial nerves problems, headache, seizures or others), presence of contrast enhancement at brain Magnetic Resonance Imaging (MRI), treatment with immunosuppressive or immunomodulant treatments or, in cases with HIV infection, treatment with combination antiretroviral therapy (cART), experimental treatments for PML, JCV-DNA levels in cerebrospinal fluid (CSF) and plasma, with distance in days from the data of diagnosis of PML, CD4 T-cell count.

For assessment of survival we considered either patients' with a date of death or with severe progression at the last observation (i.e., severe deterioration of body functions that would lead to death in a short time span) within the first year from disease onset.

MRI images were qualitatively acquired through either 1.5T or 3T equipments, based on the use of standard protocols that evolved over time. Initial protocols included at least basal axial, sagittal and coronal basal spin echo T1 and proton-density (DP)-T2-weighted sequences, with post-gadolinium T1-weighted sequences. Over time, Fluid Attenuated Inversion Recovery (FLAIR) and Diffusion Weighted Imaging (DWI) sequences were added to most of the protocols. Images were initially acquired on 2D 5 mm-thick sections, and, during most recent periods, by volumetric sequences, such as 3D-FLAIR, which enable standard 5mm-thick section reconstruction.

Quantitative analysis of JCV-DNA in CSF and plasma was performed in the first sample available since the time of diagnosis, by a real-time PCR developed in our laboratory, with a lower detection limit of 100 copies/mL.

Peripheral blood CD4+ T lymphocytes counts were determined by flow cytometry, whereas HIV-RNA was measured in plasma by commercially available assays with a detection limit of 50 copies/mL.

ELIGIBILITY:
Inclusion Criteria:

1. Definitive PML diagnosis by either JCV-DNA identification in the cerebrospinal fluid (CSF) or biopsy/autopsy, or a possible diagnosis based on clinico-radiological data, following revision of magnetic resonance imaging (MRI) exams by a PML expert neuroradiologist
2. Known year of PML diagnosis
3. Known underlying condition predisposing to PML development

Exclusion Criteria:

Missing all of the three above-mentioned inclusion criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with a diagnosis of PML, achieved by either JCV-DNA identification in the cerebrospinal fluid (CSF) or biopsy/autopsy, or a possible diagnosis based on clinico-radiological data, following revision of magnetic resonance imaging (MRI) exams by a PML expert neuroradiologist
Sampling Method: Probability Sample
Enrollment: 456 (Actual)
Dates: Start 1987-01-01 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
To evaluate the characteristics of PML patients over time and according to the underlying PML condition | At the time of PML diagnosis
  To evaluate the characteristics of PML patients (demographics, clinical, laboratory) over time and according to the underlying PML condition

SECONDARY OUTCOMES:
To assess PML patients' survival and associated variables | One year
  To assess PML patients' 1-year survival rates and associated variables

CONTACTS AND LOCATIONS:
Overall Officials: Paola Cinque, MD, PhD, Principal Investigator — San Raffaele Scientific institute
Locations (1):
- San Raffaele Scientific Institute, Milan, MI, Italy

IPD SHARING:
Plan to Share IPD: No